CLINICAL TRIAL: NCT00705237
Title: LUMA Lightwire Study
Brief Title: Study of the Use of LUMA Lightwire
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient findings for data analysis
Sponsor: Lahey Clinic (Other)
Responsible Party: Peter Catalano, M.D., Lahey Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCID 2007-118
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Sinusitis
Keywords: sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Functional Endoscopic Sinus Surgery with Balloon Dilatation — Luma lightwire technology will be utilized in conjunction with fluoroscopy for patients with sinusitis undergoing functional endoscopic sinus surgery with balloon dilatation. Trans-illumination of the sinus will be compared to fluoroscopy for accuracy

SUMMARY:
This pilot study will evaluate the accuracy and ease of use of the LUMA light wire and whether trans-illumination of the sinuses is comparable to fluoroscopy during balloon dilation procedures.

DETAILED DESCRIPTION:
50 patients undergoing functional endoscopic with balloon dilatation sinus surgery will be studied using the light wire technology. This will be used as a guide for the surgeon to know when they are safely in the sinus by trans-illumination through the sinus wall prior to utilizing balloon dilation. Routine fluoroscopy will be used as well to verify the position of the wire, which is currently standard practice. The ease, time required, and accuracy of placement will be recorded for each case and compared to data previously collected when suing standard wire technology.

ELIGIBILITY:
Inclusion Criteria:

* patients needing endoscopic sinus surgery
* initial or previous sinus surgery subject will be included

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Time, ease and accuracy of placement - compare accuracy of trans-illumination with fluoroscopy | at conclusion of subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Catalano, M.D., Principal Investigator — Lahey Clinic Medical Center
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States